CLINICAL TRIAL: NCT03906890
Title: Chromium and Trace Element Content (Cobalt, Copper, Manganese, Molybdenum, Selenium, Vanadium, Zinc) of Pediatric Parenteral Nutrition Solutions in Canada: Are Pediatric Patients on Parenteral Nutrition Exposed to Toxic Amounts?
Brief Title: Chromium Contamination of Parenteral Nutrition
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Rare Disease Foundation Microgrant competition (Unknown)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Associate Scientist, The Hospital for Sick Children
Other Study IDs: 1000057101
Record Dates: First submitted 2019-03-21; First posted 2019-04-08 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Trace Element Excess

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It has been observed that patients on total parenteral nutrition (TPN) have high plasma chromium level. There is reason to believe that TPN solutions contain chromium and possibly other trace elements as contaminants. Chromium in particular can lead to kidney damage. The purpose of this research are 1). to collect discarded TPN samples from patients on TPN for analysis and compare analyzed concnetrations of trace elements to prescribed concentrations.

2) analyze small volume parenterals obtained from a TPN supplier for evaluation of trace elements contcentrations to be compared with what is reported on the label.

3) retrospectively collect blood levels of chromium from charts of patients on home TPN who consented to have their TPN samples analyzed (#1 above), as well as prescribed Cr in their TPN at the time blood levels are recorded.

DETAILED DESCRIPTION:
Intestinal Failure (IF) occurs when a person's gut cannot work well enough to absorb enough nutrients and fluids. In these cases, life-saving nutrition called Parenteral Nutrition (PN) is given through their veins for months or years. Unfortunately, tubes of certain nutrients that are added to PN solutions have contaminants such as chromium (Cr). While the body needs a very small amount of Cr to function properly, too much is unsafe. Patients on PN may therefore get too much Cr in the PN fluids. Too much Cr can affect kidndy function. In addition to chromium, it is also possible that other trace elements are present as contaminants. While optimal nutrition if important for growth in children, too much of any nutriteint is potenially harmful. The goals of the current study therefore are

1. Measure and compare the amount of chromium, cobalt, copper, manganese, molybdenum, selenium, vanadium and zinc in a sample of discarded PN bags versus the amount of each actually ordered in those PN bags to determine the level of contamination for each of those trace elements.
2. Compare the total delivered amounts of the above elements to the current recommended amounts for age.
3. To determine if in fact patients are receiving greater than recommended amounts of chromium and other trace elements so that decisions can be made regarding current practice at SickKids.
4. To obtain small volumePN solutions from a PN supplier for analysis of each of the above mentioned trac elements for comparios what the information listed on the label of each of those products.
5. To retrospecitvely review the charts of patients who consented to have their PN analyzed from goal #1 and record blood chromium levels done over the last 5 yrs (Jan 1/2013 - Nov 30/2018) as well as Cr content of their PN solutions at the time blood Cr levels were recorded.

All patients on PN at Sickkids were eligible to participate. Data will be collected on patients weight, age, date of birth, and PN order as well as blood levels of Cr of home PN patients for the retrspective portion of the study.

Samples will be analyzed at London Health Science Centre in their Trace Elements laboratory using a Thermo Fisher ELEMENT 2 "High Resolution Sector Field Inductively Coupled Plasma Mass Spectrometer" (HR-SF-ICP-MS). This analyzer is considered the Gold Standard of Instrumentation. Samples are assessed against NIST Traceable Standards accompanying Commercial Controls to maintain as high a degree of accuracy as possible. The report of analysis will be sent to the Principal Investigator of the study.

Statistics:

Statistical analysis will be performed on primary and derived variables using SAS. Student's t-test will be used to compare the amount of teh trace elements in the PN compared to what has been ordered. Trace elements recieved pre kg/body weight will abls be compared to the recommended amount by ASPEN.

ELIGIBILITY:
Inclusion Criteria:

* All patients on TPN followed by Sickkids

Exclusion Criteria:

* Patients not on TPN
* Patients not interested in participating.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are on TPN and are "inpatients at Sickkids" or outpatients on Home TPN.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Trace elements concentrtion in TPN | 18 months
  trace elements concentration will be measured in TPN solution using ICP-MS

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, RD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada